CLINICAL TRIAL: NCT02706171
Title: Stereotactic Radiosurgery for Soft Tissue Sarcoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: The Cooper Health System (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-073
Record Dates: First submitted 2015-10-02; First posted 2016-03-11 (Estimated); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A: pre-operative (Experimental): Radiation- CyberKnife:
  35-40 Gy over 5 fractions
  Surgery:
  Surgical resection of sarcoma
  Interventions: Radiation: CyberKnife
- B: Post-operative (Experimental): Radiation- CyberKnife:
  40 Gy over 5 fractions
  Interventions: Radiation: CyberKnife
- C: Non-resectable (Experimental): Radiation- CyberKnife:
  50 Gy over 5 fractions
  Interventions: Radiation: CyberKnife

INTERVENTIONS:
Radiation: CyberKnife
  Other Names: CK

SUMMARY:
This study is evaluating treatment with CyberKnife for soft tissue sarcomas.

DETAILED DESCRIPTION:
Because of these possible advantages of SBRT over conventional radiation, the investigators began a small pilot study to test this new treatment technique in the setting of resectable soft tissue sarcomas. The pilot study was planned for a total of 12 patients which was felt to be a good number to gauge if further expansion of this technology would be successful. As of 2/6/2015 13 participants have enrolled (two enrolled patients declined treatment on protocol and thus a total of 11 patients have been treated on protocol). As of this time, the investigators have not had seen Grade 3 or higher toxicity and no instance of local failure. There have been several distant failures which would not be related to local therapy like SBRT and if anything, SBRT should reduce instance of distant failure by shortening time to chemotherapy.

The following represents the initial experience for SBRT for STS (from manuscript submitted for publication). Note that on the below abstract 8 participants were treated on the pilot study while 5 participants were treated prior to pilot study opening (the one instance of local failure is from patient treated pre-protocol).

In terms of patient numbers the goal is to have 33 patients in cohorts one and two. Using historical controls of late toxicity rates of 40% and late toxicity rates in the initial population of 20% with an alpha of 0.1 (which is reasonable for phase II studies, an alpha of 0.05 is typical for phase III studies) there would be 80% power to detect a difference with 33 patients.

The expectation for this phase II study includes the following

1. Late toxicity 30% or less
2. Local control rates 90% or better

These numbers are based on historical controls and previous research. Local control rates for historical series have been 90% or better and this also held true in the initial phase II study. For late toxicity rates, historical controls are 35-43% (The NCI study that used similar wound complication definitions to us and was a well powered study had a wound complication rate of 43%). The investigators feel that for this study to be promising enough for large phase III non-inferiority studies that the current phase II study should have late toxicity rates of 30% or better and local control rates of 90% or better.

ELIGIBILITY:
Inclusion Criteria:

* All cohorts:
* Age > 18
* Patients of child-bearing age must agree to contraception until radiosurgery has been completed.
* Note that patients with metastatic disease are eligible for protocol
* Cohort 1: Soft tissue sarcoma (of any histology subtype) in patients that are -planned to have pre-operative radiation followed by surgical resection
* Anatomical site to include upper extremity (including shoulder) and lower extremity (including hip)
* Patient performance status and co-morbid conditions to allow for surgical resection
* Cohort 2: soft tissue sarcoma (of any histologic subtype) post-resection with no further plans for additional surgery.
* Patients must have high risk feature requiring post-operative radiation which can include Large tumor (> 5 cm), High grade, Previous unplanned, non, oncologic surgery, Close margins
* Anatomical site to include upper extremity (including shoulder) and lower extremity (including hip)
* Cohort 3: soft tissue sarcoma (of any histologic subtype) that is not amenable to surgical resection for any reason
* Anatomical site to include upper extremity (including shoulder) and lower extremity (including hip and pelvis)
* Patients cannot have planned surgical resection
* Note that retroperitoneal sarcomas are not eligible

Exclusion Criteria:

-Tumors that do not fit criteria for any of the above cohorts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1-2 months
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1 year
Progression Free Survival | 5 years

SECONDARY OUTCOMES:
change in tumor burden by RECIST 1.1 response assessment | 1-2 months, 4 months
overall survival | 6 months, 1 year, 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- MD Anderson Cancer Center at Cooper, Camden, New Jersey, United States

REFERENCES:
- [Derived] Kubicek GJ, Kim TW, Gutowski CJ, Kaden M, Eastwick G, Khrizman P, Xu Q, Lackman R. Preoperative Stereotactic Body Radiation Therapy for Soft-Tissue Sarcoma: Results of Phase 2 Study. Adv Radiat Oncol. 2021 Nov 20;7(2):100855. doi: 10.1016/j.adro.2021.100855. eCollection 2022 Mar-Apr. PMID 35387414